CLINICAL TRIAL: NCT02253186
Title: Monocentre, Controlled, Randomized, Open Label, Clinical Study to Assess Safety and Efficacy of Auto-Adjustable MOBIDERM(R) Arm Sleeve in the Management of Upper Limb Lymphoedema During Night-time of Maintenance Phase
Brief Title: Clinical Study to Assess Safety and Efficacy of a New Armsleeve in the Management of Arm Lymphoedema
Acronym: MARILYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A01008-39
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Experimental): Patients wear, for 90 days, the experimental Auto-Adjustable MOBIDERM® Armsleeve during night-time and a usual custom-made compressive armsleeve during Day-time.
  Interventions: Device: Auto-Adjustable MOBIDERM Armsleeve
- Group II (No Intervention): Patients wear, for 30 days, only a usual custom-made compressive armsleeve during Day-time and no garment during night-time. Then, for the next 60 days, patients wear the experimental Auto-Adjustable MOBIDERM® Armsleeve during night-time and a usual custom-made compressive armsleeve during Day-time.

INTERVENTIONS:
Device: Auto-Adjustable MOBIDERM Armsleeve
  Other Names: MOBIDERM Autofit
  Arms: Group I

SUMMARY:
The objective of the study is to assess the effect of a new Armsleeve, worn during the night during maintenance phase of upper limb lymphoedema treatment in combination with Day-time usual lymphology hosiery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral secondary upper limb lymphoedema of stage II or III, following breast cancer
* Patients hospitalized for an intensive phase of decongestive lymphoedema therapy (DLT) for whom a decrease of lymphoedema volume has been achieved during hospitalization
* Lymphoedema with evident pitting sign (assessed as ++ or +++)
* Requiring compression therapy for, at least, the next 3 months.
* Affected arm that fits with one of the 6 standard sizes of the Auto-Adjustable MOBIDERM® armsleeve provided.
* Signed informed consent prior to any study-mandated procedure.
* Not under any administrative or legal supervision.
* Covered by a health insurance system

Exclusion Criteria:

* Stage I lymphoedema
* Active cellulitis
* Lymphoedema associated with active cancer needing acute chemotherapy
* Motor and sensitive neurological deficiency
* Post-operative oedema (i.e acute oedema following breast cancer-related surgery)
* Patient participating in any other clinical study
* Unlikely to be followed up to 3 months with clinical assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in excess arm volume | between Day 0 and Day 30
  Excess arm volume is defined as the volumetric difference between the affected upper limb compared to the contralateral upper limb, calculated with truncated cone formula

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Quere, Prof, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier - Hôpital St Eloi - Service Maladies Vasculaires, Montpellier, France